CLINICAL TRIAL: NCT03210142
Title: Minimally Invasive Hypoglossal Nerve Stimulation Study
Brief Title: Minimally Invasive Hypoglossal Nerve Stimulation Study (Lingual Study)
Acronym: Lingual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MDT16057
Record Dates: First submitted 2017-06-14; First posted 2017-07-06 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep Apnea, Neural Stimulation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transvenous hypoglossal nerve stimulation (Experimental): Transvenous hypoglossal nerve stimulation for subjects undergoing an EP, cardiac catheterization or device procedure.
  Interventions: Procedure: Transvenous hypoglossal nerve stimulation

INTERVENTIONS:
Procedure: Transvenous hypoglossal nerve stimulation — Transvenous hypoglossal nerve stimulation to open upper airway.

SUMMARY:
The purpose of this study is to assess the effect of Transvenous Hypoglossal Nerve Stimulation (tHGNS) on tongue position in the upper airway. Activation of the HGN will cause contraction of the genioglossus muscle, which will move the tongue forward, opening the upper-airway and reducing apnea-hypopnea events in patients with Obstructive Sleep Apnea (OSA). A transvenous approach will be less risky and traumatic than current HGNS systems that require an open surgical approach to wrap a cuff electrode around the HGN.

DETAILED DESCRIPTION:
The primary objective is to determine the effect of tHGNS on tongue position in the upper airway in subjects undergoing an EP, cardiac catheterization or device procedure. (Measured as changes in the anteroposterior dimensions (2-dimensional) of the retropalatal and retrolingual airway spaces.) This will be an acute study lasting no more than 45 min during a standard new device implant, cardiac catheterization and/or EP procedure. The hypoglossal nerve will be stimulated from the lingual vein using various stimulation parameters. Tongue motion, upper airway opening or any side effects will be recorded. At the end of the test procedure all hardware - the catheters, lead and/or guide wire will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old
* Subject is undergoing a standard new device implant, cardiac catheterization involving right heart catheterization and/or EP procedures
* Subject is able and willing to give informed consent

Exclusion Criteria:

* Subject is unable or unwilling to participate with study procedures
* Subject is pregnant (all women with childbearing potential must have a negative pregnancy test within 7 days prior to enrollment)
* Subject is known to be allergic to radio opaque dye
* Subject has a body mass index (BMI) >40 kg/m2
* Subject has had prior neck surgery that may interfere with vascular access to the lingual vein
* Subject has had prior surgery of the oral cavity that may interfere with tongue or soft palate movement
* Subject has a significant upper airway-related anatomic anomaly
* Subject is enrolled in a concurrent study that may confound the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Effect of transvenous hypoglossal nerve stimulation on tongue position | During study procedure
  Measured in changes in the anteroposterior dimensions (2-dimensional) of the retropalatal and retrolingual airway spaces from lateral fluoroscopic images.

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong (3):
  - Grantham Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No